CLINICAL TRIAL: NCT03906734
Title: Alfieri Stich Versus Secondary Cord Cutting During Septal Myectomy in Patients With Hypertrophic Obstructive Cardiomyopathy: A Pilot Randomized Trial
Brief Title: Mitral Valve Management During Septal Myectomy
Acronym: MVMSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01-12-3.1
Record Dates: First submitted 2019-01-20; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: septal myectomy; hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alfieri technique + Septal myectomy (Experimental): Septal myectomy plus mitral valve repair using alfieri stich
  Interventions: Procedure: Septal myectomy; Procedure: alfieri stich
- Subvalvular intervention + Septal myectomy (Active Comparator): Septal myectomy plus subvalvular mitral valve intervention
  Interventions: Procedure: Septal myectomy; Procedure: Subvalvular intervention

INTERVENTIONS:
Procedure: Septal myectomy — Transaortic septal myectomy
Procedure: alfieri stich — Transaortic Mitral valve repair using alfieri technique
  Arms: alfieri technique + Septal myectomy
Procedure: Subvalvular intervention — Transaortic Mitral valve subvalvular intervention including anterior mitral leaflet secondary cord cutting, papillary muscle release
  Arms: Subvalvular intervention + Septal myectomy

SUMMARY:
Objective of the study: to evaluate whether alfieri technique improves clinical and hemodynamic results compared to transaortic mitral valve secondary cord cutting in patients scheduled to septal myectomy for severely symptomatic hypertrophic obstructive cardiomyopathy.

DETAILED DESCRIPTION:
There is pilot prospective randomised study comparing immediate and early results of additional subvalvular mitral apparatus intervention versus additional alfieri stich in patients scheduled to septal myectomy for symptomatic obstructive cardiomyopathy.

Patients with proven hypertrophic cardiomyopathy and resting left ventricle outflow tract obstruction underwent septal myectomy. If patients were suitable for both surgical techniques, they were randomized to alfieri stich or secondary cord cutting. All surgeons were experienced at least 50 related procedures.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic obstructive cardiomyopathy
* Left ventricle outflow tract gradient > 50 mm Hg at rest
* Systolic anterior motion mediated mitral regurgitation

Exclusion Criteria:

* Intrinsic valvular heart disease
* Coronary artery disease
* Aortic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Transmitral pressure gradient | 30-days
  Transmitral pressure gradient after the procedures assessed by echocardiography

SECONDARY OUTCOMES:
Repeat bypass | 30 day
  Rate of second cross clamping and repeating bypass for procedure related reasons
Residual left ventricle outflow tract gradient | intraoperative measuerment
  Residual left ventricle outflow tract gradient assessed by direct measurement
Early mortality | 30 days
  All cause death during 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No
Restricted by local policy